CLINICAL TRIAL: NCT06449625
Title: Semaglutide Treatment for PRevention Of Toxicity in High-dose Chemotherapy With Autologous Haematopoietic Stem Cell Transplantation
Brief Title: Semaglutide in Auto-HSCT
Acronym: PROTECT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Klaus Gottlob Müller (Other)
Collaborators: Novo Nordisk A/S (Industry); Independent Research Fund Denmark (Industry)
Responsible Party: Sponsor-Investigator, Klaus Gottlob Müller, Professor, consultant, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: U1111-1277-7868; 2022-502139-20-00 (EU CTIS Number)
Record Dates: First submitted 2024-05-14; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Intestinal Mucositis; Inflammation; Chemotherapeutic Toxicity
Keywords: Gut epithelial barrier; Chemotherapy-induced toxicity; Growth factor
MeSH Terms: conditions — Inflammation | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: randomized 1:1
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide (Active Comparator): Semaglutide active drug 0.25-0.5mg, once-weekly, injection
  Interventions: Drug: Semaglutide Pen Injector [Ozempic]
- Placebo (Placebo Comparator): Semaglutide placebo, once-weekly, injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide Pen Injector [Ozempic] — Semaglutide active drug
  Arms: Semaglutide
Drug: Placebo — semaglutide placebo
  Arms: Placebo

SUMMARY:
The primary objective of this clinical trial is to ievaluate the effect of semaglutide (GLP-1 receptor agonist) in reducing intensity of gastrointestinal (GI) mucositis in patients undergoing high-dosage chemotherapy followed by autologous (auto) haematopoietic stem cell transplantation (HSCT). The secondary objective is to evaluate the effect and safety of semaglutide in reducing gut barrier injury and systemic inflammation in patients undergoing auto-HSCT.

Study design:

The study is designed as a randomized, double-blind, placebo-controlled, phase 2, two-centre investigator-initiated clinical study.

Patients referred for treatment with high-dose chemotherapy and auto-HSCT will be randomized in a 1:1 manner to receive either semaglutide or placebo. The study includes a run-in period 3 to 4-week low-dose period with semaglutide subcutaneously (s.c.) 0.25 mg once-weekly (QW) prior to high-dose chemotherapy treatment followed by a period of 4 to 5 weeks with semaglutide 0.5 mg QW. Total duration of treatment with investigational drug will be 8 weeks. Total study duration for the individual patients will be 20-22 weeks, including a 2-4-week screening period and 10 weeks of follow-up.

Study population:

A planned total number of 40 patients will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Referral for auto-HSCT for relapsed diffuse large B-cell lymphoma or follicular lymphoma
* Age ≥ 18 years
* BMI ≥ 18.5
* ECOG performance status* ≤ 2
* Literate in Danish and/or English

Exclusion Criteria:

* Diabetes
* Inflammatory bowel disease
* Previous or current gastrointestinal malignancy
* Personal or family history of medullary thyroid carcinoma or MEN syndrome
* Genetic disorders with defective tissue repair (e.g., Fanconi anaemia)
* History of pancreatitis (acute or chronic)
* Renal impairment measured as eGFR value of < 30 ml/min/1.73 m2
* Impaired liver function, defined as alanine aminotransferase ≥ 2.5 times upper normal limit at screening
* Known or suspected hypersensitivity to semaglutide or other GLP-1RA
* Pregnant or nursing females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-12 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
gastrointestinal mucositis severity | from day of stem cell infusion (day 0) to week +3
  mean severity grade (0-II)

SECONDARY OUTCOMES:
CRP increment | from day of stem cell infusion (day 0) to week +3
  AUC
Quality of life general | change from baseline (start of high-dose chemotherapy) to study week 9 and 18
  evaluated by EORTC QLQ-C30 questionnaire. The QLQ-C30 summary score is calculated as the mean of the combined 13 QLQ-C30 scale and item scores (excluding global QoL and financial impact). Final scoring range: 0-100 with a higher score indicating a better quality of life
Quality of life - high-dose chemotherapy treatment specific | change from baseline (start of high-dose chemotherapy) to study week 9 and 18
  evaluated by EORTC QLQ-HDC29 questionnaire. The QLQ HDC29 module includes 29 items, consisting of 6 multi-item scales and 8 singleitems. Final scoring range: 0-100 with a higher score indicating a better quality of life
Safety profile evaluated by number of SARs | Start of study drug treatment (week 1) until study week 10
  SAR will be estimated according to ICH-GCP guidelines

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sorum ME, Gang AO, Tholstrup DM, Gudbrandsdottir S, Kissow H, Kornblit B, Muller K, Knop FK. Semaglutide treatment for PRevention Of Toxicity in high-dosE Chemotherapy with autologous haematopoietic stem-cell Transplantation (PROTECT): study protocol for a randomised, double-blind, placebo-controlled, investigator-initiated study. BMJ Open. 2024 Oct 9;14(10):e089862. doi: 10.1136/bmjopen-2024-089862. PMID 39384243